CLINICAL TRIAL: NCT04486924
Title: Evaluation of the Acute Performance and Safety of the Globe® Mapping and Ablation System With the GPS™ Module for the Treatment of Atrial Fibrillation
Brief Title: Performance and Safety of the Globe® Mapping and Ablation System With the GPS™ Module for the Treatment of Atrial Fibrillation
Acronym: GPS-CA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kardium Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: DOC-150565
Record Dates: First submitted 2020-07-22; First posted 2020-07-27 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Globe Mapping and Ablation System (Experimental)
  Interventions: Device: Globe Mapping and Ablation System

INTERVENTIONS:
Device: Globe Mapping and Ablation System — Prospective, non-randomized, open-label clinical study.

SUMMARY:
This study will evaluate the safety and acute performance of the Globe® Mapping and Ablation System with the GPS™ Module intended to conduct electroanatomic mapping and ablation treatment of subjects with atrial fibrillation (AF).

ELIGIBILITY:
Inclusion Criteria:

1. ≥18 years old and ≤75 years old
2. Symptomatic AF with at least one AF episode electrocardiographically documented within one (1) year prior to enrolment. Documentation may include diagnosis in the patient medical files, electrocardiogram (ECG), Trans-telephonic monitoring (TTM), Holter monitor or telemetry strip.
3. Selected for catheter ablation for the treatment of atrial fibrillation

Exclusion Criteria:

1. History of previous left atrial ablation or surgical treatment for AF/AFL/AT
2. Contraindication for either catheter ablation or epicardial surgery (including, but not limited to: previous thoracic radiation, previous perimyocarditis, previous cardiac tamponade, pleural adhesions, and prior thoracotomy)
3. Presence of LA thrombus by TEE, CT scan, MRI, or angiography
4. Known conditions or anatomical abnormality that may interfere with the device delivery or positioning (e.g. myxoma, tumour, calcification, venous access path narrowing, or tortuosity)
5. Planned concomitant cardiac surgery procedures besides AF treatment (valve, coronary, others)
6. Uncontrolled heart failure or NYHA Class III or IV heart failure
7. Valve repair or replacement or presence of a prosthetic valve
8. Coronary artery bypass grafting, cardiac surgery, or valvular cardiac surgical procedure within the past 6 months
9. MI or PCI procedure within 3 months before screening
10. Left Ventricular Ejection Fraction (LVEF) < 40%
11. Presence of implanted pacemaker or implantable cardioverter defibrillator (ICD)
12. Severe pulmonary hypertension or prior pulmonary stenting
13. History of cerebrovascular disease, including stroke or transient ischemic attack (TIA) within 6 months prior to enrollment
14. Contraindication to anticoagulation (e.g., heparin)
15. History of blood clotting or bleeding disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2021-04-05 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
Acute isolation of all clinically relevant pulmonary veins confirmed by entrance block | start to end of the procedure
Procedure time | start to end of the procedure
Catheter dwell time | start to end of the procedure
Fluoroscopy time | start to end of the procedure
Fluoroscopy dose area product | start to end of the procedure
Incidence of Primary Adverse Events (PAE) occurring peri-procedurally and within 7 days (inclusive) of the ablation procedure | start to seven days after the end of the procedure
Incidence of all serious adverse events occurring peri-procedurally and within 7 days (inclusive) of the ablation procedure | start to seven days after the end of the procedure

CONTACTS AND LOCATIONS:
Overall Officials: Southlake Regional Health Centre, Principal Investigator — 596 Davis Dr, Newmarket ON L3Y 2P9, Canada
Locations (2):
- Canada (2):
  - Southlake Regional Health Centre, Newmarket
  - St. Paul's Hospital, Vancouver